CLINICAL TRIAL: NCT00126581
Title: A Phase II Randomized Study of OSI-774 (Erlotinib) (NSC #718781) With or Without Carboplatin/Paclitaxel in Patients With Previously Untreated Adenocarcinoma of the Lung Who Never Smoked or Were Former Light Smokers
Brief Title: Erlotinib Hydrochloride With or Without Carboplatin and Paclitaxel in Treating Patients With Stage III-IV Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00464; NCI-2009-00464 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000437097; CALGB-30406 (Other: Alliance for Clinical Trials in Oncology); CALGB-30406 (Other: CTEP); U10CA180821 (NIH); U10CA031946 (NIH)
Record Dates: First submitted 2005-08-02; First posted 2005-08-04 (Estimated); Results first posted 2014-04-23 (Estimated); Last update posted 2019-08-07 (Actual); Status verified 2019-07

CONDITIONS: Lung Adenocarcinoma; Lung Adenosquamous Carcinoma; Malignant Pericardial Effusion; Malignant Pleural Effusion; Minimally Invasive Lung Adenocarcinoma; Stage IIIB Lung Non-Small Cell Cancer AJCC v7; Stage IV Lung Non-Small Cell Cancer AJCC v7
Keywords: A Phase II Randomized Study of OSI-774
MeSH Terms: conditions — Adenocarcinoma of Lung; Pleural Effusion, Malignant; Adenocarcinoma, Bronchiolo-Alveolar | interventions — Carboplatin; Erlotinib Hydrochloride; Paclitaxel; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (erlotinib hydrochloride) (Experimental): Patients receive erlotinib hydrochloride PO QD on days 1-21. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Erlotinib; Drug: Erlotinib Hydrochloride
- Arm II (erlotinib hydrochloride, paclitaxel, carboplatin) (Experimental): Patients receive erlotinib hydrochloride as in arm I. Patients also receive paclitaxel IV over 1-3 hours and carboplatin IV over 15-30 minutes on day 1. Treatment repeats every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. After completion of 6 cycles of treatment, patients may continue to receive erlotinib hydrochloride alone as above.
  Interventions: Drug: Carboplatin; Drug: Erlotinib; Drug: Erlotinib Hydrochloride; Drug: Paclitaxel

INTERVENTIONS:
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
  Arms: Arm II (erlotinib hydrochloride, paclitaxel, carboplatin)
Drug: Erlotinib — Given PO
Drug: Erlotinib Hydrochloride — Given PO
  Other Names: Cp-358,774; OSI-774; Tarceva
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
  Arms: Arm II (erlotinib hydrochloride, paclitaxel, carboplatin)

SUMMARY:
This randomized phase II trial studies how well erlotinib hydrochloride with or without carboplatin and paclitaxel works in treating patients with stage III-IV non-small cell lung cancer. Erlotinib hydrochloride may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as carboplatin and paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving erlotinib hydrochloride together with carboplatin and paclitaxel may kill more tumor cells than giving either drug alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the distribution of progression-free survival (PFS) in patients with previously untreated advanced adenocarcinoma of the lung who are never or light former smokers treated with either OSI-774 (erlotinib) (erlotinib hydrochloride) alone (arm A) or in combination with carboplatin/paclitaxel (arm B).

SECONDARY OBJECTIVES:

I. To determine the radiographic response rate in patients with previously untreated advanced adenocarcinoma of the lung who are never or light former smokers treated with either OSI-774 (erlotinib) alone (arm A) or in combination with carboplatin/paclitaxel (arm B).

II. To determine the frequency of epidermal growth factor receptor (EGFR) and V-Ki-ras2 Kirsten rat sarcoma viral oncogene homolog (K-ras) mutations and anaplastic lymphoma kinase (ALK) translocations in patients with previously untreated advanced adenocarcinoma of the lung who are never or light former smokers.

III. To determine the response rate and time to progression in patients with and without EGFR mutations treated with either OSI-774 (erlotinib) alone (arm A) or in combination with carboplatin/paclitaxel (arm B).

IV. To determine the response rate and time to progression in patients with and without K-ras mutations treated with either OSI-774 (erlotinib) alone (arm A) or in combination with carboplatin/paclitaxel (arm B).

V. To determine the median and overall survival of patients with previously untreated advanced adenocarcinoma of the lung who are never or light former smokers treated with either OSI-774 (erlotinib) alone (arm A) or in combination with carboplatin/paclitaxel (arm B).

VI. To estimate the response rate, progression-free, and overall survival of patients with echinoderm microtubule associated protein like (EML)4-ALK translocation who received OSI-774 erlotinib alone (arm A) or in combination with carboplatin/paclitaxel (arm B).

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive erlotinib hydrochloride orally (PO) once daily (QD) on days 1-21. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive erlotinib hydrochloride as in Arm I. Patients also receive paclitaxel intravenously (IV) over 1-3 hours and carboplatin IV over 15-30 minutes on day 1. Treatment repeats every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. After completion of 6 cycles of treatment, patients may continue to receive erlotinib hydrochloride alone as above.

After completion of study treatment, patients are followed at least every 3 months for 1 year and then every 6 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologic documentation of primary lung adenocarcinoma including any variant thereof such as pure or mixed bronchioloalveolar carcinoma or adenosquamous cell carcinoma; patients with non-small cell lung cancer (NSCLC) not otherwise specified (NOS) are not eligible

  * Pathology block or unstained slides from initial or subsequent diagnosis must be available for sequencing of EGFR, K-ras, Erb-2 and B-raf; patients need to have had at least a core biopsy; patients whose diagnosis was made through a fine needle aspirate will not have sufficient material for mutational analysis and are not eligible
* Select stage IIIB with cytologically documented malignant pleural or pericardial effusion OR stage IV disease
* Patients must be chemotherapy naïve; they may not have received neo-adjuvant or adjuvant chemotherapy
* No prior exposure to OSI-774 (erlotinib) or other treatments targeting the human epidermal growth factor receptor (HER) family axis (e.g., trastuzumab, gefitinib, cetuximab, lapatinib, etc.)
* No uncontrolled central nervous system metastases (i.e., any known central nervous system [CNS] lesion which is radiographically unstable, symptomatic and/or requiring corticosteroids); patients must be >= 3 weeks beyond completing cranial irradiation and off corticosteroid therapy
* >= 3 weeks since prior radiation therapy
* >= 3 weeks since prior major surgery
* No treatment with an investigational agent currently or within the last 28 days
* Non-smoker or former light smoker; non-smoker is defined as a person who smoked =< 100 cigarettes in their lifetime while a former light smoker is a patient who smoked between > 100 cigarettes AND =< 10 pack years AND quit >= 1 year ago; this must be documented on the On-study Form (C-1405)
* Eastern Cooperative Oncology Group (ECOG) 0 or 1
* Non-pregnant and non-nursing
* No dysphagia or active gastrointestinal disease or disorder that alters gastrointestinal motility or absorption; no lack of integrity of the gastrointestinal tract (e.g., a significant surgical resection of the stomach or small bowel); patients unable to swallow intact tablets must be able to swallow tablets dissolved in water
* Measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 20 mm with conventional techniques or as >= 10 mm with spiral computed tomography (CT) scan; lesions that are considered non-measurable include the following:

  * Bone lesions
  * Leptomeningeal disease
  * Ascites
  * Pleural/pericardial effusion
  * Lymphangitis cutis/pulmonis
  * Abdominal masses that are not confirmed and followed by imaging techniques
  * Cystic lesions
* Granulocyte >= 1,500/mcl
* Platelet count >= 100,000/mcl
* Hemoglobin >= 9.0 g/dL
* Total bilirubin =< upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) =< 2.5 x ULN
* Creatinine =< 1.5 mg/dl

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2005-08-15 (Actual); Primary Completion 2010-06-30 (Actual); Study Completion 2017-11-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pasi A Janne, Principal Investigator — Alliance for Clinical Trials in Oncology
Locations (96):
- United States (96):
  - East Bay Radiation Oncology Center, Castro Valley, California
  - Eden Hospital Medical Center, Castro Valley, California
  - Valley Medical Oncology Consultants-Castro Valley, Castro Valley, California
  - Bay Area Breast Surgeons Inc, Emeryville, California
  - Valley Medical Oncology Consultants-Fremont, Fremont, California
  - Saint Rose Hospital, Hayward, California
  - Contra Costa Regional Medical Center, Martinez, California
  - El Camino Hospital, Mountain View, California
  - Highland General Hospital, Oakland, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Tumor Institute, Oakland, California
  - Hematology and Oncology Associates-Oakland, Oakland, California
  - Tom K Lee Inc, Oakland, California
  - Valley Care Health System - Pleasanton, Pleasanton, California
  - Valley Medical Oncology Consultants, Pleasanton, California
  - University of California San Diego, San Diego, California
  - Kaiser Permanente-San Diego Mission, San Diego, California
  - Veterans Administration-San Diego Medical Center, San Diego, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - Doctors Medical Center- JC Robinson Regional Cancer Center, San Pablo, California
  - Middlesex Hospital, Middletown, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Jupiter Medical Center, Jupiter, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Memorial Health University Medical Center, Savannah, Georgia
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - AMITA Health Adventist Medical Center, La Grange, Illinois
  - Elkhart General Hospital, Elkhart, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - IU Health La Porte Hospital, La Porte, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - MedStar Franklin Square Medical Center/Weinberg Cancer Institute, Baltimore, Maryland
  - Union Hospital of Cecil County, Elkton, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mass General/North Shore Cancer Center, Danvers, Massachusetts
  - Cape Cod Hospital, Hyannis, Massachusetts
  - Lowell General Hospital, Lowell, Massachusetts
  - South Shore Hospital, South Weymouth, Massachusetts
  - Lakeland Medical Center Saint Joseph, Saint Joseph, Michigan
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Missouri Cancer Associates, Columbia, Missouri
  - Veterans Administration, Columbia, Missouri
  - University of Missouri - Ellis Fischel, Columbia, Missouri
  - Capital Region Medical Center, Jefferson City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Center for Cancer Care and Research, St Louis, Missouri
  - CHI Health Saint Francis, Grand Island, Nebraska
  - Great Plains Health Callahan Cancer Center, North Platte, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Saint Joseph Hospital, Nashua, New Hampshire
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Hematology Oncology Associates of Central New York-East Syracuse, East Syracuse, New York
  - Northwell Health NCORP, Lake Success, New York
  - North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Ralph Lauren Center for Cancer Care and Prevention, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Saint Joseph's Hospital Health Center, Syracuse, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Wayne Radiation Oncology, Goldsboro, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - Vidant Oncology-Kinston, Kinston, North Carolina
  - Wilson Medical Center, Wilson, North Carolina
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Cancer Care Associates, Oklahoma City, Oklahoma
  - Memorial Hospital of Rhode Island, Pawtucket, Rhode Island
  - Rhode Island Hospital, Providence, Rhode Island
  - Miriam Hospital, Providence, Rhode Island
  - Roper Hospital, Charleston, South Carolina
  - McLeod Regional Medical Center, Florence, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Greenville Memorial Hospital, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Eastside, Greenville, South Carolina
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - Rappahannock General Hospital, Kilmarnock, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between August 2005 and April 2009, 188 participants were enrolled.
Pre-assignment Details: Seven participants withdrew consent before initiating study therapy, therefore, 181 participants were randomized to either arm.
Groups:
- Arm A: Erlotinib: Patients receive oral erlotinib once daily on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
- Arm B: Erlotinib/Carboplatin/Paclitaxel: Patients receive erlotinib as in arm I. Patients also receive paclitaxel IV over 1-3 hours and carboplatin IV over 15-30 minutes on day 1. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. After completion of 6 courses of treatment, patients may continue to receive erlotinib alone as above.
Period: Overall Study
Arm/Group | Arm A: Erlotinib | Arm B: Erlotinib/Carboplatin/Paclitaxel
Started | 81 | 100
Completed | 68 | 80
Not Completed | 13 | 20
Not completed — Adverse Event | 3 | 7
Not completed — Death | 3 | 2
Not completed — Withdrawal by Subject | 1 | 4
Not completed — Alternative therapy | 3 | 3
Not completed — Other illness/MD discretion | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Erlotinib | Arm B: Erlotinib/Carboplatin/Paclitaxel | Total
Number analyzed (Participants) | 81 | 100 | 181
Age, Continuous [Median (Full Range); unit: years] | 58 [32 to 78] | 60 [34 to 81] | 59 [32 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 58 | 107
  Male | 32 | 42 | 74
Region of Enrollment [Number; unit: participants]
  United States | 81 | 100 | 181
ECOG Performance Status [Number; unit: participants] — Classifies patients according to their functional impairment. Scores range from 0 (fully active) to 5 (death).
  participants
    0 - fully active | 50 | 48 | 98
    1 - minimal symptoms | 31 | 52 | 83
Smoking history [Number; unit: participants]
  Never smoker | 64 | 79 | 143
  Light former smoker | 17 | 21 | 38
Histology [Number; unit: participants]
  Adenocarcinoma | 71 | 84 | 155
  Bronhioloalveolar cancer | 2 | 2 | 4
  Adenocarcinoma with bronchioloalveolar features | 8 | 14 | 22

OUTCOME MEASURES:

1. Primary Outcome: 18 Weeks Progression Free Survival (PFS) Rate
Description: The product limit estimator developed by Kaplan Meier will be used to graphically describe progression free survival for patients randomized to each study arm.
  The 18 week progression-free survival rate was defined as the proportion of patients that were alive progression-free 18 weeks after registration into the study. Disease progression was assessed per modified RECIST criteria, and defined as at least a 20% increase in the sum of the longest diameters of target lesions, in either primary or nodal lesions, taking as reference the smallest sum longest diameter recorded since the baseline measurements, or the appearance of new lesions. Kaplan-Meier estimate of 18-week progression-free survival was calculated.
Time Frame: At 18 weeks
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: Erlotinib | Arm B: Erlotinib/Carboplatin/Paclitaxel
Number analyzed (Participants) | 81 | 100
percentage of participants | 52 [NA to NA] — The 80% Confidence Interval was computed = (45, 59). | 69 [NA to NA] — The 80% Confidence Interval was computed = (62, 74).

2. Secondary Outcome: Overall Response Rate
Description: The proportion of patients who respond (completely or partially) to each combination regimen will be estimated. An exact binomial confidence interval will be computed for these estimates.
  Response was defined using Response Evaluation Criteria In Solid Tumors (RECIST) criteria:
  Complete Response (CR): disappearance of all target lesions; Partial Response (PR) 30% decrease in sum of longest diameter of target lesions
Time Frame: Duration of Study (up to 3 years)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: Erlotinib | Arm B: Erlotinib/Carboplatin/Paclitaxel
Number analyzed (Participants) | 81 | 100
percentage of participants | 35 [24 to 46] | 46 [36 to 56]

3. Secondary Outcome: Number of Participants With Grade 3, 4 or 5 Adverse Event at Least Possibly Related to Treatment.
Description: The National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 3.
  Grade 1: Mild; Grade 2: Moderate; Grade 3: Severe; Grade 4: Life Threatening; Grade 5: Death.
Time Frame: Duration of study (up to 3 years)
Measure: Number; unit: participants
Arm/Group | Arm A: Erlotinib | Arm B: Erlotinib/Carboplatin/Paclitaxel
Number analyzed (Participants) | 81 | 99
participants | 20 | 52

4. Other Pre Specified Outcome: Overall Survival
Description: Overall survival (OS) is defined as the time from patient randomization (arm assignment) to death from any cause. The median OS with 95% CI was estimated using the Kaplan-Meier method.
Time Frame: Time from randomization to death (up to 3 years)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Erlotinib | Arm B: Erlotinib/Carboplatin/Paclitaxel
Number analyzed (Participants) | 81 | 100
months | 24.6 [18.4 to 33.8] | 19.8 [14.4 to 27.8]

5. Other Pre Specified Outcome: Progression Free Survival (PFS) by Epidermal Growth Factor Receptor (EGFR) Mutation Status
Description: PFS was defined as the time from registration until disease progression or death, whichever occurs first. The median PFS with 95% CI was estimated using the Kaplan-Meier method. Progression is defined as in the primary outcome measure.
  EGFR mutations were performed at the Dana-Farber Cancer Institute using a sensitive heteroduplex method coupled with enzymatic digestion as previously reported (Janne PA, et al: A rapid and sensitive enzymatic method for epidermal growth factor receptor mutation screening. Clin Cancer Res 12:751-758, 2006). All positive findings were independently verified and subjected to sequencing. The mutation analyses were blinded to the participants' clinical outcome.
Time Frame: Duration of treatment (up to 3 years)
Population: EGFR mutation analysis was successfully performed in 164 participants; 17 participants had insufficient material or DNA for analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Erlotinib | Arm B: Erlotinib/Carboplatin/Paclitaxel
Number analyzed (Participants) | 77 | 87
months
  EGFR Mutant | 14.1 [7.0 to 19.6] | 17.2 [8.2 to 28.7]
  EGFR Wild Type | 2.6 [1.4 to 3.9] | 4.8 [2.8 to 5.6]

6. Other Pre Specified Outcome: Overall Response Rate by EGFR Mutation Status
Description: Response and EGFR mutation status are defined in previous outcome measures.
Time Frame: Duration of study (up to 3 years)
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Arm A: Erlotinib | Arm B: Erlotinib/Carboplatin/Paclitaxel
Number analyzed (Participants) | 77 | 87
percentage of participants
  EGFR Mutant | 70 [51 to 84] | 73 [18 to 44]
  EGFR Wild Type | 9 [3 to 22] | 30 [18 to 44]

7. Other Pre Specified Outcome: Progression Free Survival With KRAS Mutation Status
Description: Progression free survival is defined in previous outcome measures. GIven the small number of KRAS mutant participants, the analysis combines data from both arms.
Time Frame: Duration of study (up to 3 years)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Mutant | Wild Type
Number analyzed (Participants) | 17 | 147
months | 4 [2.8 to 12.4] | 6.7 [5.3 to 8.0]

8. Other Pre Specified Outcome: Overall Response Rate With KRAS Mutational Status
Description: Overall response is defined in previous outcome measures. GIven the small number of KRAS mutant participants in each treatment arm, the analysis combines data from both arms.
Time Frame: Duration of study (up to 3 years)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Mutant | Wild Type
Number analyzed (Participants) | 17 | 147
percentage of participants | 29 [10 to 56] | 42 [34 to 51]

ADVERSE EVENTS:
Arm/Group | Arm A: Erlotinib | Arm B: Erlotinib/Carboplatin/Paclitaxel
Serious Adverse Events (participants affected / at risk) | 21/81 | 39/99
Other Adverse Events (participants affected / at risk) | 78/81 | 94/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Erlotinib (N=81) | Arm B: Erlotinib/Carboplatin/Paclitaxel (N=99)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 8 (9)
Hemoglobin (Blood and lymphatic system disorders) | 9 (10) | 20 (25)
Hemolysis (e.g. immune hemolytic anemia drug-related hemolysis) (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac Arrhythmia - Other (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac General - Other (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac ischemia/infarction (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 2 (2)
Vision-blurred vision (Eye disorders) | 0 (0) | 1 (1)
Watery eye (epiphora tearing) (Eye disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (3) | 7 (9)
Diarrhea (Gastrointestinal disorders) | 8 (9) | 20 (26)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 2 (2)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 2 (3) | 3 (5)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 3 (4)
Hemorrhage, GI (Gastrointestinal disorders) | 2 (2) | 4 (5)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 2 (2)
Mucositis/stomatitis (clinical exam) (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mucositis/stomatitis (functional/symptomatic) (Gastrointestinal disorders) | 2 (3) | 4 (4)
Nausea (Gastrointestinal disorders) | 5 (5) | 21 (25)
Pain (Gastrointestinal disorders) | 6 (6) | 6 (6)
Ulcer GI (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 5 (5) | 12 (14)
Death not associated with CTCAE term (General disorders) | 3 (3) | 1 (1)
Edema: limb (General disorders) | 4 (4) | 3 (3)
Edema: viscera (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 10 (12) | 25 (34)
Fever (General disorders) | 4 (4) | 6 (6)
Pain - Other (General disorders) | 1 (1) | 1 (1)
Rigors/chills (General disorders) | 2 (2) | 3 (3)
Gallbladder pain (Hepatobiliary disorders) | 0 (0) | 1 (1)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 2 (2) | 3 (3)
Infection with normal ANC or Grade 1 or 2 neutrophils (Infections and infestations) | 2 (2) | 5 (5)
Infection with unknown ANC (Infections and infestations) | 2 (2) | 1 (1)
Bruising (in absence of Grade 3 or 4 thrombocytopenia) (Injury, poisoning and procedural complications) | 1 (2) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 3 (3)
Alanine aminotransferase increased (Investigations) | 2 (2) | 5 (6)
Alkaline phosphatase (Investigations) | 0 (0) | 2 (2)
Amylase (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 5 (5) | 8 (11)
Blood bilirubin increased (Investigations) | 4 (4) | 7 (9)
CPK (creatine phosphokinase) (Investigations) | 1 (1) | 0 (0)
Creatinine (Investigations) | 1 (1) | 7 (8)
INR (International Normalized Ratio of prothrombin time) (Investigations) | 2 (2) | 6 (8)
Leukocytes (total WBC) (Investigations) | 1 (1) | 24 (25)
Lipase increased (Investigations) | 1 (1) | 0 (0)
Lymphopenia (Investigations) | 2 (2) | 9 (13)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 0 (0) | 19 (19)
Platelet count decreased (Investigations) | 2 (2) | 14 (18)
Weight loss (Investigations) | 2 (2) | 4 (4)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 6 (6) | 10 (13)
Anorexia (Metabolism and nutrition disorders) | 7 (8) | 13 (17)
Bicarbonate, serum-low (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Calcium serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 2 (2) | 1 (2)
Calcium serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 1 (1) | 9 (11)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 9 (9)
Glucose serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 1 (1) | 12 (15)
Glucose serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Magnesium serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 1 (1) | 8 (12)
Phosphate serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 0 (0) | 4 (5)
Potassium serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 1 (1) | 4 (4)
Potassium serum-low (hypokalemia) (Metabolism and nutrition disorders) | 2 (2) | 6 (8)
Sodium serum-high (hypernatremia) (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Sodium serum-low (hyponatremia) (Metabolism and nutrition disorders) | 3 (3) | 11 (11)
Triglyceride serum-high (hypertriglyceridemia) (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Arthritis (non-septic) (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Muscle weakness, generalized or specific area (not due to neuropathy) (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (2) | 7 (9)
Headache (Nervous system disorders) | 2 (2) | 2 (2)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 1 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2) | 20 (30)
Speech impairment (e.g., dysphasia or aphasia) (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 2 (2) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2)
Confusion (Psychiatric disorders) | 0 (0) | 3 (3)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (3) | 4 (5)
Cystitis (Renal and urinary disorders) | 0 (0) | 1 (1)
Glomerular filtration rate (Renal and urinary disorders) | 0 (0) | 1 (1)
Hemoglobinuria (Renal and urinary disorders) | 0 (0) | 2 (2)
Hemorrhage GU (Renal and urinary disorders) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1) | 2 (3)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary frequency/urgency (Renal and urinary disorders) | 1 (2) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Adult Respiratory Distress Syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Allergic rhinitis (including sneezing nasal stuffiness postnasal drip) (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Bronchospasm wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 10 (12)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 12 (14)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Obstruction/stenosis of airway (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary/Upper Respiratory - Other (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Voice changes/dysarthria (e.g. hoarseness loss or alteration in voice laryngitis) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (2) | 13 (18)
Dermatology/Skin - Other (Skin and subcutaneous tissue disorders) | 2 (3) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4)
Nail changes (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 2 (2) | 9 (10)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 15 (16) | 16 (22)
Flushing (Vascular disorders) | 1 (1) | 0 (0)
Hemorrhage/Bleeding - Other (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 2 (3)
Hypotension (Vascular disorders) | 0 (0) | 3 (3)
Thrombosis/thrombus/embolism (Vascular disorders) | 3 (3) | 9 (9)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Erlotinib (N=81) | Arm B: Erlotinib/Carboplatin/Paclitaxel (N=99)
Blood/Bone Marrow - Other (Blood and lymphatic system disorders) | 1 (7) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 6 (6)
Hemoglobin (Blood and lymphatic system disorders) | 19 (89) | 62 (357)
Hemolysis (e.g. immune hemolytic anemia drug-related hemolysis) (Blood and lymphatic system disorders) | 0 (0) | 5 (7)
Palpitations (Cardiac disorders) | 2 (4) | 2 (2)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 2 (2)
Supraventricular and nodal arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (4) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 2 (3)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 1 (3)
Otitis external ear (non-infectious) (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (8) | 5 (8)
Endocrine - Other (Endocrine disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 2 (8) | 2 (9)
Cataract (Eye disorders) | 2 (2) | 1 (1)
Conjunctivitis (Eye disorders) | 0 (0) | 3 (6)
Dry eye syndrome (Eye disorders) | 8 (30) | 5 (54)
Eye pain (Eye disorders) | 2 (2) | 0 (0)
Eyelid dysfunction (Eye disorders) | 2 (4) | 3 (4)
Keratitis (Eye disorders) | 2 (30) | 0 (0)
Ocular/Visual - Other (Eye disorders) | 3 (6) | 3 (12)
Ophthalmoplegia/diplopia (double vision) (Eye disorders) | 0 (0) | 2 (2)
Photophobia (Eye disorders) | 3 (21) | 1 (1)
Retinopathy (Eye disorders) | 1 (2) | 0 (0)
Vision-blurred vision (Eye disorders) | 4 (6) | 6 (12)
Vision-flashing lights/floaters (Eye disorders) | 1 (1) | 0 (0)
Watery eye (epiphora tearing) (Eye disorders) | 1 (4) | 2 (11)
Abdominal distension (Gastrointestinal disorders) | 1 (4) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 2 (4)
Constipation (Gastrointestinal disorders) | 16 (99) | 34 (97)
Dental: teeth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 66 (480) | 76 (401)
Dry mouth (Gastrointestinal disorders) | 7 (42) | 9 (68)
Dyspepsia (Gastrointestinal disorders) | 17 (68) | 18 (60)
Dysphagia (Gastrointestinal disorders) | 4 (4) | 11 (15)
Flatulence (Gastrointestinal disorders) | 2 (5) | 1 (1)
Gastritis (including bile reflux gastritis) (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal - Other (Gastrointestinal disorders) | 3 (6) | 1 (2)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 1 (2)
Hemorrhage, GI (Gastrointestinal disorders) | 2 (12) | 3 (5)
Hemorrhoids (Gastrointestinal disorders) | 2 (4) | 4 (6)
Mucositis/stomatitis (clinical exam) (Gastrointestinal disorders) | 5 (15) | 11 (18)
Mucositis/stomatitis (functional/symptomatic) (Gastrointestinal disorders) | 13 (109) | 16 (37)
Nausea (Gastrointestinal disorders) | 33 (127) | 53 (156)
Oral pain (Gastrointestinal disorders) | 6 (15) | 3 (4)
Pain (Gastrointestinal disorders) | 16 (65) | 24 (84)
Salivary gland changes/saliva (Gastrointestinal disorders) | 2 (6) | 0 (0)
Stricture/stenosis (including anastomotic) GI (Gastrointestinal disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Typhlitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 12 (18) | 27 (50)
Constitutional Symptoms - Other (General disorders) | 1 (12) | 2 (2)
Death not associated with CTCAE term (General disorders) | 4 (7) | 1 (1)
Edema: limb (General disorders) | 9 (39) | 12 (26)
Edema:head and neck (General disorders) | 2 (3) | 0 (0)
Facial pain (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 44 (350) | 79 (528)
Fever (General disorders) | 6 (6) | 8 (11)
Flu-like syndrome (General disorders) | 0 (0) | 2 (2)
Injection site reaction/extravasation changes (General disorders) | 0 (0) | 1 (5)
Pain - Other (General disorders) | 7 (28) | 8 (17)
Rigors/chills (General disorders) | 6 (6) | 3 (11)
Syndromes - Other (General disorders) | 0 (0) | 3 (5)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Gallbladder pain (Hepatobiliary disorders) | 1 (1) | 2 (5)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 3 (6) | 14 (20)
Autoimmune reaction (Immune system disorders) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 12 (26) | 17 (31)
Infection - Other (Infections and infestations) | 4 (6) | 5 (15)
Infection with normal ANC or Grade 1 or 2 neutrophils (Infections and infestations) | 14 (40) | 13 (53)
Infection with unknown ANC (Infections and infestations) | 3 (6) | 5 (7)
Infection without neutropenia (Infections and infestations) | 2 (2) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Prostate infection (Infections and infestations) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 1 (3) | 1 (7)
Bruising (in absence of Grade 3 or 4 thrombocytopenia) (Injury, poisoning and procedural complications) | 2 (43) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (4)
Intra-operative injury (Injury, poisoning and procedural complications) | 1 (4) | 0 (0)
Rash: dermatitis associated with radiation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thrombosis/embolism (vascular access-related) (Injury, poisoning and procedural complications) | 0 (0) | 2 (3)
Vessel injury-vein (Injury, poisoning and procedural complications) | 0 (0) | 1 (4)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 19 (50) | 18 (48)
Alkaline phosphatase (Investigations) | 13 (31) | 19 (65)
Amylase (Investigations) | 0 (0) | 1 (5)
Aspartate aminotransferase increased (Investigations) | 18 (74) | 39 (91)
Blood bilirubin increased (Investigations) | 19 (137) | 32 (214)
Cholesterol serum-high (hypercholesteremia) (Investigations) | 1 (1) | 0 (0)
Creatinine (Investigations) | 13 (45) | 18 (119)
GGT (gamma-Glutamyl transpeptidase) (Investigations) | 1 (1) | 0 (0)
Haptoglobin (Investigations) | 0 (0) | 1 (2)
INR (International Normalized Ratio of prothrombin time) (Investigations) | 1 (1) | 12 (21)
Leukocytes (total WBC) (Investigations) | 10 (56) | 63 (259)
Lipase increased (Investigations) | 0 (0) | 1 (5)
Lymphopenia (Investigations) | 8 (72) | 18 (69)
Metabolic/Laboratory - Other (Investigations) | 1 (3) | 3 (6)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 2 (11) | 45 (117)
Platelet count decreased (Investigations) | 5 (62) | 43 (123)
Weight loss (Investigations) | 3 (4) | 13 (29)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 15 (46) | 25 (115)
Anorexia (Metabolism and nutrition disorders) | 31 (94) | 35 (120)
Bicarbonate, serum-low (Metabolism and nutrition disorders) | 0 (0) | 2 (5)
Calcium serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 4 (24) | 2 (2)
Calcium serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 6 (10) | 15 (27)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 7 (14)
Glucose serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 15 (41) | 33 (105)
Glucose serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 0 (0) | 5 (5)
Magnesium serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 1 (1) | 1 (2)
Magnesium serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 7 (14) | 18 (77)
Phosphate serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 1 (2) | 3 (3)
Potassium serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 11 (33) | 7 (10)
Potassium serum-low (hypokalemia) (Metabolism and nutrition disorders) | 16 (31) | 20 (60)
Sodium serum-high (hypernatremia) (Metabolism and nutrition disorders) | 1 (1) | 5 (5)
Sodium serum-low (hyponatremia) (Metabolism and nutrition disorders) | 6 (19) | 17 (47)
Triglyceride serum-high (hypertriglyceridemia) (Metabolism and nutrition disorders) | 0 (0) | 1 (14)
Arthralgia (Musculoskeletal and connective tissue disorders) | 16 (107) | 21 (88)
Arthritis (non-septic) (Musculoskeletal and connective tissue disorders) | 2 (11) | 2 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 12 (35) | 16 (91)
Bone pain (Musculoskeletal and connective tissue disorders) | 10 (46) | 10 (18)
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 8 (26) | 9 (15)
Joint-function (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (5)
Muscle weakness, generalized or specific area (not due to neuropathy) (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (3)
Musculoskeletal/Soft Tissue - Other (Musculoskeletal and connective tissue disorders) | 2 (3) | 7 (13)
Myalgia (Musculoskeletal and connective tissue disorders) | 10 (51) | 21 (39)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (9) | 4 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 (36) | 14 (33)
Secondary Malignancy - possibly related to cancer treatment (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 0 (0) | 3 (7)
Depressed level of consciousness (Nervous system disorders) | 1 (3) | 0 (0)
Dizziness (Nervous system disorders) | 10 (25) | 17 (28)
Dysgeusia (Nervous system disorders) | 10 (58) | 23 (84)
Extrapyramidal disorder (Nervous system disorders) | 1 (14) | 0 (0)
Headache (Nervous system disorders) | 12 (65) | 12 (28)
Laryngeal nerve dysfunction (Nervous system disorders) | 0 (0) | 1 (2)
Memory impairment (Nervous system disorders) | 1 (2) | 2 (2)
Neurology - Other (Nervous system disorders) | 0 (0) | 2 (7)
Neuropathy: cranial (Nervous system disorders) | 0 (0) | 2 (2)
Peripheral motor neuropathy (Nervous system disorders) | 3 (10) | 4 (8)
Peripheral sensory neuropathy (Nervous system disorders) | 18 (78) | 58 (632)
Seizure (Nervous system disorders) | 1 (2) | 1 (2)
Sinus pain (Nervous system disorders) | 0 (0) | 1 (1)
Speech impairment (e.g., dysphasia or aphasia) (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Vasovagal episode (Nervous system disorders) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 2 (3)
Anxiety (Psychiatric disorders) | 14 (53) | 8 (53)
Confusion (Psychiatric disorders) | 2 (5) | 3 (3)
Depression (Psychiatric disorders) | 5 (25) | 11 (49)
Insomnia (Psychiatric disorders) | 17 (99) | 24 (85)
Personality change (Psychiatric disorders) | 0 (0) | 1 (1)
Glomerular filtration rate (Renal and urinary disorders) | 0 (0) | 1 (1)
Hemoglobinuria (Renal and urinary disorders) | 0 (0) | 1 (4)
Hemorrhage GU (Renal and urinary disorders) | 0 (0) | 2 (2)
Obstruction, GU (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal/Genitourinary - Other (Renal and urinary disorders) | 2 (3) | 3 (4)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 1 (3)
Urinary frequency/urgency (Renal and urinary disorders) | 2 (25) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (2) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Ejaculatory dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (2)
Irregular menses (change from baseline) (Reproductive system and breast disorders) | 0 (0) | 2 (3)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 2 (3)
Vaginal dryness (Reproductive system and breast disorders) | 1 (4) | 0 (0)
Allergic rhinitis (including sneezing nasal stuffiness postnasal drip) (Respiratory, thoracic and mediastinal disorders) | 10 (73) | 9 (38)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchospasm wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 2 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 44 (174) | 45 (142)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 31 (158) | 35 (92)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9 (29) | 10 (21)
Hemorrhage pulmonary/upper respiratory (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Nasal cavity/paranasal sinus reactions (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (7)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 6 (7)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (8)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 3 (8) | 2 (2)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (2)
Pulmonary/Upper Respiratory - Other (Respiratory, thoracic and mediastinal disorders) | 7 (29) | 5 (31)
Voice changes/dysarthria (e.g. hoarseness loss or alteration in voice laryngitis) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 7 (10)
Alopecia (Skin and subcutaneous tissue disorders) | 18 (103) | 58 (325)
Dermatology/Skin - Other (Skin and subcutaneous tissue disorders) | 11 (46) | 11 (65)
Dry skin (Skin and subcutaneous tissue disorders) | 25 (232) | 29 (144)
Nail changes (Skin and subcutaneous tissue disorders) | 13 (80) | 11 (113)
Pain of skin (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (1)
Photosensitivity (Skin and subcutaneous tissue disorders) | 2 (4) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 10 (99) | 11 (32)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 24 (131) | 42 (180)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 69 (632) | 73 (806)
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 3 (27) | 4 (5)
Skin breakdown/decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Sweating (diaphoresis) (Skin and subcutaneous tissue disorders) | 3 (4) | 0 (0)
Ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (4)
Flushing (Vascular disorders) | 1 (1) | 0 (0)
Hematoma (Vascular disorders) | 0 (0) | 1 (1)
Hemorrhage/Bleeding - Other (Vascular disorders) | 1 (2) | 3 (12)
Hot flashes/flushes (Vascular disorders) | 1 (1) | 2 (4)
Hypertension (Vascular disorders) | 8 (97) | 7 (35)
Hypotension (Vascular disorders) | 0 (0) | 3 (3)
Phlebitis (including superficial thrombosis) (Vascular disorders) | 0 (0) | 2 (4)
Thrombosis/thrombus/embolism (Vascular disorders) | 3 (3) | 3 (5)
Vascular - Other (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less